CLINICAL TRIAL: NCT04743973
Title: A Feasibility Study Evaluating Mindfulness-Based Intervention Assessing A Wearable Wellness Brain Sensing Device (Muse-S) in Practicing Physicians
Brief Title: A Study to Asses Wellness Using a Brain Sensing Device on Physicians
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: InteraXon, Inc. (Industry); Cambridge Brain Sciences (Industry)
Responsible Party: Principal Investigator, Ivana T Croghan, PhD, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-007207
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Results first posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Stress, Emotional; Sleep; Quality of Life
Keywords: mindfulness; Wellness
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Practicing Physicians (Experimental): Practicing physicians at Mayo Clinic caring for patients during the COVID 19 pandemic will receive the Muse S™ Headband system, and will be asked to utilize it at least 4 times per week for a minimum of 10 minutes each time over a period of 3 months (12 weeks).
  Interventions: Device: Muse S™ Headband system

INTERVENTIONS:
Device: Muse S™ Headband system — Brain sensing headband that measures brain activity by detecting electrical impulses created by the brain.

SUMMARY:
A study to asses the feasibility of physicians using a wearable brain sensing wellness device during a time of increased work load, patient volume and stressors to assess the association between duration of active state and calm state as measured by the wearable brain sensing wellness device, and quality of life (QOL), subjective stress, sleep and resilience.

DETAILED DESCRIPTION:
Participants will be instructed on how to use a brain sensing device and corresponding digital application to engage in structured digital mindfulness practices daily for 3 months. Subjects will be requested to use the device and practice daily, but the amount of time and frequency daily will be to their choosing. Subjects will also complete questionnaires and cognitive based testing throughout participation.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older at time of consent
* Practicing Physicians at Mayo Clinic
* Not pregnant by subject self-report at time of consent
* Have the ability to provide informed consent
* Have the ability to complete all aspects of this trial
* Have access to a smart phone or tablet device
* Have no contraindicating comorbid health condition which would interfere with the proper use of the Muse-S™ system, as determined by the clinical investigators

Exclusion Criteria:

* Used an investigational drug within the past 30 days
* Currently (within the past 3 weeks) been practicing mindfulness training on a weekly/regular basis
* Currently (within 3 weeks) been enrolled in another clinical or research program (e.g. CAM) which intervenes on the patients' QOL, or stress
* An unstable medical or mental health condition as determined by the physician investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-08-15 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivana T Croghan, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ghosh K, Nanda S, Hurt RT, Schroeder DR, West CP, Fischer KM, Bauer BA, Fokken SC, Ganesh R, Hanson JL, Lindeen SA, Pruthi S, Croghan IT. Mindfulness Using a Wearable Brain Sensing Device for Health Care Professionals During a Pandemic: A Pilot Program. J Prim Care Community Health. 2023 Jan-Dec;14:21501319231162308. doi: 10.1177/21501319231162308. PMID 36960553

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who were patients in the long COVID-19 clinic were invited to participate if they were found to be eligible for the study.
Groups:
- Muse-S Group: Participants used Muse-S for the study period (up to 3 months).
Period: Overall Study
Arm/Group | Muse-S Group
Started | 40
Completed | 35
Not Completed | 5
Not completed — Withdrawal by Subject | 5

BASELINE CHARACTERISTICS:
Arm/Group | Muse-S Group
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] — Age in years at baseline.
  years | 41.3 (11.0)
Sex: Female, Male [Count of Participants; unit: Participants] — Sex of participant at birth
  Participants
    Female | 34
    Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Hispanic or Latino Ethnicity that is self-identified by participants
  Participants
    Hispanic or Latino | 2
    Not Hispanic or Latino | 38
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Self-identified race by participants
  Participants
    American Indian or Alaska Native | 0
    Asian | 2
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 1
    White | 35
    More than one race | 1
    Unknown or Not Reported | 1
Perceived Stress Scale baseline score [Mean (Standard Deviation); unit: units on a scale] — The Perceived Stress Scale (PSS) is a 10-item Likert scale that measures global life stress by assessing the degree to which experiences are appraised as uncontrollable or unpredictable. Scores can range from 0 to 40, with higher scores indicating greater perceived stress.
  units on a scale | 11.1 (3.94)
Resilience baseline score [Mean (Standard Deviation); unit: units on a scale] — Resilience was measured using the Connor-Davison Resilience Scale 10 (CD-RS10). This is a 10-item, likert scale, validated, scoring system. With the higher score indicating higher resilience. The CD-RS10 is a reliable means of assessing resilience and most often used in medical and/or disaster studies
  units on a scale | 27.4 (5.01)
LASA baseline score [Mean (Standard Deviation); unit: units on a scale] — Quality of Life was measured using the validated Linear Analogue Self-Assessment (LASA) scale. This measure is a six-item measure of quality of life (QOL), in which QOL is conceptualized as a multidimensional construct with five domains (physical, functional, emotional, spiritual, and social). This is a 11-item Likert scale (0 to 10) with 0 being the worst possible and 10 being the best possible.
  units on a scale | 39.2 (6.59)

OUTCOME MEASURES:

1. Primary Outcome: Frequency Adherence to Intervention
Description: Summarizing frequency subjects use intervention during active study participation (during 3 month study period)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: times used
Arm/Group | Muse-S Group
Number analyzed (Participants) | 40
times used | 57.8 (30.6)

2. Primary Outcome: Duration Adherence to Intervention
Description: Summarizing duration of time subjects use intervention during active study participation (during 3 month time period)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Muse-S Group
Number analyzed (Participants) | 40
minutes | 5.9 (1.9)

3. Secondary Outcome: Perceived Stress Scale (PSS) Score Difference
Description: The Perceived Stress Scale (PSS) is a 10-item 5-point Likert scale that measures global life stress by assessing the degree (Never, almost never, sometimes, often and very often) to which experiences are appraised as uncontrollable or unpredictable. Scores can range from 0 to 40, with higher scores indicating greater perceived stress. The score difference is the average change from Day 90 to Baseline.
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Muse-S Group
Number analyzed (Participants) | 36
units on a scale | -2.1 (3.81)

4. Secondary Outcome: Resilience Score Difference
Description: Resilience was measured using the Connor-Davison Resilience Scale 10 (CD-RS10). This is a 10-item, 5-point likert scale, validated, scoring system. Scores can range from 0 to 40, with higher scores indicating higher resilience. The CD-RS10 is a reliable means of assessing resilience and most often used in medical and/or disaster studies. Difference from Day 90 to baseline for the resilience score
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Muse-S Group
Number analyzed (Participants) | 36
units on a scale | 1.4 (3.9)

5. Secondary Outcome: LASA Score Difference
Description: Quality of Life was measured using the validated Linear Analogue Self-Assessment (LASA) scale. This measure is a 6-item, 11-point likert scale, validated scoring system that measure of quality of life (QOL), in which QOL is conceptualized as a multidimensional construct with five domains (physical, functional, emotional, spiritual, and social). In this measure, each domain can score 0 as the worst possible and 10 being the best possible. The total score for QoL could range from 0 to 60 with higher score indicating greater QoL. Change from Day 90 to Baseline for the LASA score
Time Frame: 90 days
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Muse-S Group
Number analyzed (Participants) | 36
units on a scale | 2.7 (6.0)

ADVERSE EVENTS:
Time Frame: During the treatment phase (3 months)
Arm/Group | Muse-S Group
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 1/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Muse-S Group (N=40)
Headache (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT04743973/Prot_000.pdf
  • Statistical Analysis Plan (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/73/NCT04743973/SAP_001.pdf